CLINICAL TRIAL: NCT00869765
Title: An Open Pilot Trial of Transcranial Direct Current Stimulation (tDCS) Augmented by D-Cycloserine as a Treatment for Depression.
Brief Title: Transcranial Direct Current Stimulation (tDCS) Augmentation by D-Cycloserine as a Treatment for Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Associate Professor Colleen Loo, University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09052
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Depression; Treatment; Transcranial direct current stimulation; D-cycloserine
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression | interventions — Cycloserine; Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tDCS and D-CYC (Experimental): Major Depression tDCS and D-cyc
  Interventions: Drug: D-Cycloserine; Device: tDCS (Eldith DC-Stimulator (CE certified))

INTERVENTIONS:
Drug: D-Cycloserine — 100 mg D-cycloserine once every weekday taken 2 hours before tDCS session.
Device: tDCS (Eldith DC-Stimulator (CE certified)) — tDCS session lasting continuously for 20 minutes at 2 mA. Conductive rubber electrodes (7 x 5 cm, 35 cm2) covered by sponges soaked in saline will be used, held in place by a head band. The current will be gradually increased to the level of 2 mA over 30 seconds (to avoid the sensation of a flash).
  Other Names: Eldith DC-Stimulator (CE certified)

SUMMARY:
Among antidepressant treatments, Electroconvulsive therapy (ECT) stands as the most effective in treating acute depression. However, patient concerns with the cognitive side effects of ECT have encouraged the development of new and more focal forms of brain stimulation such as transcranial Direct Current Stimulation (tDCS). The investigators' current study of tDCS as a treatment for depression suggests that this technique has antidepressant effects and is safe, painless and well tolerated. However, not all patients may respond to this treatment and the concern of possible relapse in some patients who respond to tDCS has raised interest in finding treatments that may enhance and prolong the antidepressant effects of tDCS. This study will investigate whether D-Cycloserine, a medication shown to lengthen the effects of tDCS on brain activity, can also enhance/prolong the antidepressant effects of tDCS in people suffering from depression.

ELIGIBILITY:
Inclusion Criteria:

1. Subject met inclusion criteria for study HREC 07305 (a sham controlled study of transcranial direct current stimulation (tDCS) as a treatment for depression).
2. Subject completed study HREC 07305.
3. Subject either did not reach remission at the end of trial (defined as MADRS score of ≤ 10) or suffered an early relapse (within a month of finishing the trial).

Exclusion Criteria:

1. Diagnosis (as defined by DSM-IV) of: any psychotic disorder (lifetime); bipolar disorder; eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder current or within the past year); mental retardation.
2. History of drug or alcohol abuse or dependence (as per DSM-IV criteria) within the last 3 months (except nicotine and caffeine).
3. Inadequate response to ECT in the current episode of depression.
4. Subject is on regular benzodiazepine medication which it is not clinically appropriate to discontinue.
5. Subject requires a rapid clinical response due to inanition, psychosis or high suicide risk.
6. Neurological disorder or insult, e.g., recent stroke (CVA), which places subject at risk of seizure or neuronal damage with tDCS.
7. Subject has metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
8. Female subject who is pregnant, or of child-bearing age, sexually active and not using reliable contraception (urine test for pregnancy will be used)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology (IDS-C) | 6 months

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, Principal Investigator — University of New South Wales
Locations (1):
- Black Dog Institute, University of New South Wales, Randwick, New South Wales, Australia

REFERENCES:
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au